CLINICAL TRIAL: NCT05928728
Title: The Colchicine and Atrial Fibrillation Trial
Acronym: COLFIB
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Adam Femerling Langhoff, Principal Investigator, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-500850-40-01
Record Dates: First submitted 2023-06-14; First posted 2023-07-03 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Experimental)
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Colchicine 0.5 mg once daily
  Arms: Colchicine
Drug: Placebo — Placebo once daily
  Arms: Placebo

SUMMARY:
The purpose of this study to investigate the effects of colchicine on atrial fibrillation recurrence and vascular and cardiac function in patients with atrial fibrillation.

DETAILED DESCRIPTION:
The study is an investigator-initiated, prospective, double-blind, placebo-controlled, randomized clinical trial investigating the effects of colchicine in patients with atrial fibrillation (AF). The study population will consist of approximately 500 patients aged 18 years and above with a diagnosis of paroxysmic or persistent AF with a successful outcome of cardioversion. Patients will be randomized to either low-dose colchicine treatment (0,5 mg once daily) or placebo. Treatment will continue for 12 months. Patients will be assessed by measurement of time to first admission with AF (Electro Cardio Gram (ECG) confirmed), echocardiography, cardiac Magnetic Resonance Imaging (MRI), and blood samples at baseline and after 6 + 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Living address in the Capital Region of Denmark
2. Age > 18
3. Diagnosed with paroxysmic/persistent AF.
4. Planned or acute admission for cardioversion of AF with successful outcome.
5. Female participants should either not be of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile, or is of childbearing potential and practicing one of the following methods of contraception throughout the study and for 30 days after study completion: Hormonal contraception (oral contraceptives, contraceptive implant, injectable birth control, contraceptive patch, or vaginal ring) or intrauterine device
6. Participants will have given written, informed consent and are able and willing to comply with the requirements of the study protocol.
7. Optimal background therapy (in relation to comorbidities and development of heart failure / thromboembolic event) for AF as judged by the investigator.

Exclusion Criteria:

1. Colchicine treatment for another cause, e.g. gout
2. Allergy/hypersensitivity to colchicine
3. Uncontrolled hypertension (systolic BP >180 mmHg or diastolic BP >110 mmHg)
4. History of malignancy of any organ system excluding a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma, localized prostate cancer and/or localized carcinoma in situ of the cervix
5. Cirrhosis, chronic active hepatitis or other severe hepatic disease
6. Hemodialysis
7. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2
8. Systemic treatment with moderate or strong cytochrome P450 3A4 (CYP3A4) inhibitors or P-glycoprotein inhibitors (list in Appendix 1)
9. Permanent AF
10. Female participants who are pregnant, lactating, or considering becoming pregnant during the study or for 6 months after study completion
11. Significant drug or alcohol abuse during the last year
12. Current use of or plans to initiate chronic systemic steroid therapy during the study (topical or inhaled steroids are allowed)
13. Planned ablation procedure as treatment for AF
14. If cardiovascular surgery or ablation has been done the past three months prior to inclusion.
15. Chronic inflammatory bowel disease (Crohn's disease or ulcerative colitis) or chronic diarrhea
16. Use of other investigational drugs within 30 days of the time of enrollment
17. Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
18. Suspected AF, confirmed with ECG, at time of inclusion and randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2026-06-14 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Between-group difference in change in time to first AF admission measured in days | 12 months

SECONDARY OUTCOMES:
Between-group difference in change in accumulated number of readmissions for symptomatic AF | 12 months
Between-group difference in change in Left Atrial Volume (LAV) assessed by echocardiography | 12 months
Between-group difference in change in Atrial Fibrillation Effect On Quality-Of-Life Questionnaire (AFEQT) score | 12 months
  Score of 0 being the worst outcome and score of 100 being the best outcome

OTHER OUTCOMES:
Between-group difference in change in plasma concentration of high sensitivity C-Reactive Protein (hs-CRP) | 12 months
Between-group difference in change in plasma concentration of high sensitivity Troponin I (hs-TnI) | 12 months
Between-group difference in change in Left Ventricle (LV) septal wall thickness assessed by echocardiography | 12 months
Between-group difference in change in LV mass index assessed by echocardiography | 12 months
Between-group difference in change in LV posterior wall thickness assessed by echocardiography | 12 months
Between-group difference in change in Left Ventricle Ejection Fraction (LVEF) assessed by echocardiography | 12 months
Between-group difference in change in E/A ratio assessed by echocardiography | 12 months
Between-group difference in change in e' assessed by echocardiography | 12 months
Between-group difference in change in E/e' ratio assessed by echocardiography | 12 months
Between-group difference in change in Global Longitudinal Strain (GLS) assessed by echocardiography | 12 months
Between-group difference in change in aortic distensibility assessed by echocardiography | 12 months
Between-group difference in change in aortic strain assessed by echocardiography | 12 months
Between-group difference in change in LV septal wall thickness assessed by cardiac MRI | 12 months
Between-group difference in change in LV posterior wall thickness assessed by cardiac MRI | 12 months
Between-group difference in change in LVEF assessed by cardiac MRI | 12 months
Between-group difference in change in myocardial fibrosis assessed by cardiac MRI | 12 months
Between-group difference in change in myocardial inflammation assessed by cardiac MRI | 12 months
Between-group difference in change in plasma concentration of Tumor Necrosis Factor alpha (TNF-α) | 12 months
Between-group difference in change in plasma concentration of pro Brain Natriuretic Peptide (pro-BNP) | 12 months
Between-group difference in change in accumulated number of cardiovascular-related hospital visits | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam Femerling Langhoff, M.D., Principal Investigator — Herlev and Gentofte Hospital
Locations (1):
- Center for Translational Cardiology and Pragmatic Randomized Trials (CTCPR), Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Yes